CLINICAL TRIAL: NCT06959355
Title: Examination of Frailty and Related Factors in Lumbar Spinal Stenosis
Brief Title: Frailty and Associated Factors in Lumbar Spinal Stenosis
Status: Recruiting | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Principal Investigator, PhD, Karabuk University
Other Study IDs: Karabuk-002
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with frail LSS: Patients with LSS who are frail according to Fried criteria will be assigned to this group. According to the Frid criteria, patients who score 3 or more on the following symptoms have a frailty level: weight loss, weakness, exhaustion, decreased mobility, and physical inactivity.
- Patients without frail LSS: Patients with LSS who are not frail according to Fried criteria will be assigned to this group.

SUMMARY:
Lumbar spinal stenosis (LSS) is generally seen with advanced age, but it manifests itself with an increase in both physical and psychological health problems. Frailty is an important parameter that has become increasingly important in recent years and affects both the physical and psychological health of individuals. It has been examined in various disease groups in the literature and is reported to increase in patients with low back pain. However, the level of frailty and related factors in LSS are unknown. Since physical and psychological health are important in maintaining daily life, it is important to examine frailty in these individuals who present with chronic pain symptoms.

DETAILED DESCRIPTION:
Lumbar spinal stenosis (LSS) is a degenerative disease that occurs due to compression of neurological structures as a result of narrowing of the spinal canal, and is particularly common in elderly individuals. LSS is characterized by pain, neurogenic claudication, decreased walking capacity, and functional disability. This condition can limit patients' daily living activities, leading to decreased physical activity levels, balance disorders, and increased fear of falling. At the same time, disability and decreased quality of life due to the disease can negatively affect individuals' physical and psychosocial health status, leading to increased frailty levels. Frailty is an important geriatric concept that requires multidisciplinary approaches and is associated with increased dependency and risk of falling in elderly individuals. Demonstrating the relationship between frailty and parameters such as pain, disability, quality of life, physical activity, balance, and fear of falling in individuals with LSS can contribute to the development of more effective rehabilitation strategies for the management of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lumbar spinal stenosis by MRI,
* Patients between the ages of 45-80,
* Patients who can stand independently,
* Volunteer to participate in the study

Exclusion Criteria:

* Patients who did not agree to participate in the study,
* Those with a chronic disease that would affect walking,
* Those who had undergone surgery in the lumbar region within the last year,
* Those with advanced joint disease in the lower extremity,
* Those with malignancy in the spine,
* Those with vision and/or vestibular system problems,
* Those who did not cooperate well were not included in the study.

Ages: 45 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with LSS based on magnetic resonance imaging clinical evaluation will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Pain severity | Baseline
  Pain will be assessed with the numerical pain scale (NRS). NRS varies between 0-10. The higher the score, the greater the pain.
  Pain will be assessed with the numerical pain scale (NRS). NRS varies between 0-10. The higher the score, the greater the pain.
  Pain will be assessed with the numerical pain scale (NRS). NRS varies between 0-10. The higher the score, the greater the pain.
Static balance | Baseline
  Static balance will be assessed with the one-legged standing test. The test is terminated when it is 30 seconds or more, and there is a balance disorder below 10 seconds.
  Static balance will be assessed with the one-legged standing test. The test is terminated when it is 30 seconds or more, and there is a balance disorder below 10 seconds.
Dynamic balance | Baseline
  Dynamic balance will be assessed with Timed up and Go test. Time will be recorded in seconds
Disability | Baseline
  Disability will be assessed using the Oswestry Disability Index. The scale is scored from 0 to 100. A higher score indicates greater disability.
Fear of Falling | Baseline
  Fear of falling will be assessed with the Fall Efficacy Scale-International. It is scored between 16-64, the higher the score, the greater the fear of falling.
Health related quality of life | Baseline
  Quality of life will be assessed with Short Form-36. It is scored between 0-100, the higher the score, the higher the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Gunes, PhD, Principal Investigator — Karabuk University; Aydın Sinan Apaydın, PhD, Principal Investigator — Karabuk University
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim HJ, Park S, Park SH, Lee JH, Chang BS, Lee CK, Yeom JS. The prevalence and impact of frailty in patients with symptomatic lumbar spinal stenosis. Eur Spine J. 2019 Jan;28(1):46-54. doi: 10.1007/s00586-018-5710-1. Epub 2018 Sep 1. PMID 30173327
- [Result] Leopoldino AAO, Megale RZ, Diz JBM, Moreira BS, Felicio DC, Queiroz BZ, Bastone AC, Ferreira ML, Pereira LSM. Influence of Frailty Status on Pain, Disability, and Quality of Life in Older Adults with Acute Low Back Pain: Results from the Back Complaints in the Elders (BACE-Brazil) Study. Can J Aging. 2021 Sep;40(3):367-375. doi: 10.1017/S0714980820000288. Epub 2020 Aug 14. PMID 32792030
- [Result] Nagai S, Kawabata S, Michikawa T, Ito K, Takeda H, Ikeda D, Kaneko S, Fujita N. Association between frailty and locomotive syndrome in elderly patients with lumbar spinal stenosis: A retrospective longitudinal analysis. Geriatr Gerontol Int. 2024 Jan;24(1):116-122. doi: 10.1111/ggi.14785. Epub 2023 Dec 23. PMID 38140947